CLINICAL TRIAL: NCT00281086
Title: Center for Reducing Asthma Disparities - Harvard University/Boston Area Community Health Centers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1195; U01HL072495 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-04

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

SUMMARY:
To address the problems of disparities in asthma care and morbidity by examining the influence of environmental/genetic factors and stress on the development of asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic condition affecting over 14 million Americans, but the prevalence rates are higher in certain populations (e.g. 10 percent in inner-cities and 30 percent among the homeless vs. 5 percent in a general population of whites). African Americans and Hispanics from the Northeast are twice as likely to die from asthma as whites. African Americans are four times as likely to be hospitalized for asthma and are five times more likely than whites to seek care for asthma at an emergency department. Reasons for these higher rates are not certain, and most likely result from an interaction of risk factors such as environmental exposures, genetic predisposition, access to appropriate medical care, socioeconomic status, and cultural health practices. The National Heart, Lung, and Blood Institute supports a variety of activities to address the pressing public health problems posed by asthma. However, progress in reducing disparities has been disappointingly slow. Separate, independent research projects have generated important clues for understanding the nature and scope of the problem. A more coordinated, interdisciplinary and comprehensive approach to research is needed to take advantage of these clues, move the science further and faster, and increase our capacity to improve health outcomes among minority and economically disadvantaged populations. Cooperative centers of research that foster partnerships among minority medical centers, research intensive institutions, and the communities in which asthma patients live will promote such advancement.

The Request for Applications for the Centers for Reducing Asthma Disparities was released in October, 2001. The objective of the program is to promote partnerships (called Centers) between a minority serving institution (MSI) that may not have a strong research program and a research intensive institution (RII) that has a track record of NIH-supported research and patient care. The purpose of the partnership is to conduct collaborative research on asthma disparities (i.e. greater prevalence of asthma, higher rates of morbidity due to asthma, and lesser access or use of quality medical care among minorities and poor).

DESIGN NARRATIVE:

The Center for Reducing Asthma Disparities involves partnership between researchers at Harvard University (Channing Laboratory, Brigham and Women's Hospital, and the Harvard School of Public Health) and a network of Boston-area Community Health Centers (CHCs) affiliated with the non-profit community-based organization CCHERS (Center for Community Health Education, Research and Service). Broad specific aims are: 1. Conduct a community needs assessment to assess differences in perceptions about asthma etiology, disparities, and effective treatment between community representatives, Community Health Center patients, and Community Health Center providers. 2. Determine the role of socio/environmental exposures (psychosocial stress, indoor allergens, cigarette smoking and diesel-related air pollutants) on asthma onset through study of a prenatally enrolled birth cohort. 3. Determine the role of genetics in modifying the risk of the social/physical environment by concurrent assessment of the following genetic factors thought to influence immune development and airway inflammation in early life: stress (corticosteroid regulatory genes, adrenergic system regulatory genes), diesel exhaust and smoking (biotransformation genes), indoor allergens (cytokine pathway genes). 4. Use a quasi-experimental design to evaluate the effectiveness of the research, training, and outreach components of the project in leading to significant changes in the ability of particular stakeholders to design and implement sound asthma intervention strategies. 5. Develop training programs at Harvard that provide masters and predoctoral students as well as postdoctoral fellows with experience and expertise in Community-Based Participatory Research (CBPR) focused on reducing asthma disparities. 6. Develop training and information dissemination materials for health center staff and community members (especially caregivers of children with asthma). The Center for Community Health Education, Research and Service will take the lead in implementing Specific Aims 1, 4 and 6, while the Harvard group will take the lead on Aims 2, 3 and 5. In addition to building needed infrastructure to support partnership-based research and interventions aimed at reducing health disparities, this proposal has the potential to make significant contributions to the scientific literature with respect to health disparities and asthma.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Piltch — Center for Community Health Education Research & Service; Rosalind Wright — Brigham and Women's Hospital